CLINICAL TRIAL: NCT06017388
Title: A Neurophenomenological Study of Hypnosis
Brief Title: Mystical Experience in Hypnosis: a Neurophenomenological Study
Acronym: MystHyp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bicego Aminata, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-213
Record Dates: First submitted 2023-08-02; First posted 2023-08-30 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Healthy
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The control group will simply receive a reading of the mystical experience suggestion without hypnosis.
  Interventions: Behavioral: Control
- Experiemental (Experimental): The experiemental group will receive a suggestion of the mystical experience in hypnosis.
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — We will propose a hypnotic induction followed by a suggestion of mystical experience (based on Lynn & Evans, 2017).
  Arms: Experiemental
Behavioral: Control — We will propose the neutral reading of a mystical expetience suggestion (based on Lynn & Evans, 2017).
  Arms: Control

SUMMARY:
Mystical experience is described as an experience that is unique to everyone, potentially transformative and leaving a mark for many years or even a lifetime. It is characterized by: a loss of self/ego, being with the whole/nature/universe, transcendence, a loss of spatio-temporal reference points, ineffability, peace and joy, a sacred character, and a noetic quality. The mystical experience is one that occurs in the context of non-ordinary states of consciousness such as meditation and the consumption of so-called psychedelic drugs, for example. It would seem, in fact, to correspond to the transformative mechanism of the psychedelic experience. The goal ofthis study is to investigate the possibility of a mystical experience through hypnosis.

DETAILED DESCRIPTION:
Anyone interested in taking part in the study will be contacted by telephone or e-mail and offered a face-to-face appointment to carry out the screening (T0). During the appointment, screening (cf. inclusion criteria) will be carried out, socio-demographic data (age, sex, education, nationality, history of hypnosis practice, etc.) and randomization will also take place at this time. At this time, the investigators will assess psychological flexibility and psychologigal well-being, and participants will do a cognitive flexibility task (T1). If people meet the inclusion criteria, the investigators will schedule an appointment for a session to take place roughly a week later.

During this session, the investigators will start by reviewing beliefs about hypnosis, assessing participants' expectations of the study, their absorption and dissociation trait, their positive and negative affects and their anxiety. Next, the investigators will perform a 15-minute resting electroencephalographic (EEG) recording. We will then administer the Elkins Hypnotizability Scale. A 30-minute break will be taken. Next, the investigators willperform a hypnotic induction followed by a mystical experience suggestion for the experimental group. The control group will simply receive a reading of the mystical experience suggestion without hypnosis. The rest of the procedure is the same for both groups. EEG activity will be recorded during the mystical experience suggestion (± 15 minutes) in hypnosis and outside hypnosis (ordinary state of consciousness). Directly afterwards, participants will be asked to orally explain their subjective experience during the suggestion of mystical experience. Then the investigators will assess the positive and negative affect in addition to these outcomes: the mystical experience, the ego dissolution, the psychological flexibility, the cognitive flexibility, the altered state of consciousness, the near-death experience, alterness, absorption state, dissociation state, time perception (T2).

Three months after receiving the experimental session, participants will be seen again for a follow-up session (T3). During this session, we will ask: "Since the experimental session, have you observed any changes in your behaviors, emotions and beliefs? If so, can you tell us about them?". The investigators will assess the positive and negative affects and psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* good comprehension of French

Exclusion Criteria:

* Psychiatric history
* History of neurological disorder
* Psychoactive medication
* Addiction
* Alcoholism

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Mystical experience | During the procedure
  The 30-item revised Mystical Experience Questionnaire will assess the occurrence and intensity of mystical-type experiences. It is comprised of four factors: mysticality, positivity of mood, transcendence of time and space, and ineffability. A mystical experience is defined as having a score equal or above 60% on all factors.
Hypnotizability | During the procedure
  The susceptibility one has concerning hypnosis. Will be assessed with the Elkins Hypnotizability Scale. A score :
  0-3 : low hypnotizability 4-7: medium hypnotizability 8-11 : high hypnotizability 12 : very high hypnotizability.

SECONDARY OUTCOMES:
Ego Dissolution | During the procedure
  The Ego Dissolution Inventory will assess the occurrence of ego dissolution.
Alteration of consciousness | During the procedure
  The Phenomenology of Consciousness Inventory will allow to empirically quantify the subjective experience in terms of pattern and intensity parameters. It is composed of 53 items consisting of 12 major dimensions (e.g., positive affect), and 14 minor dimensions (e.g., absorption) (annex). Graphs will be constructed to represent the intensity and pattern of relationships between pairs of dimensions.
Psychological flexibility | Before the procedure and direclty after the procedure
  Multidimensional Psychological Flexibility Inventory.
Cognitive flexibility | Before the procedure and direclty after the procedure
  Cognitive flexility will be assessed with the Test of Attentional Performance which is an informatized cognitive task.
Psychological well-being | Before the intervention and after 3 months
  Psychological well-being will be assessed with the Warwick-Edinburgh Mental Well-Being Scale
Modification of mood, cognition, emotion and behavior | After 3 months
  We will ask an open-ended question "Since the experimental session, have you observed any changes in your behaviors, emotions and beliefs? If so, can you tell us about them?".
Phenomenal experience | During the procedure
  Phenomenal experience will be assessed by the recording of the narrative experience.

OTHER OUTCOMES:
Socio-demographics | At screening
  age, sex, éducation, nationality, prior practice of hypnosis or other non-ordinary states of consciousness, prior mystical experience.
Psychiatric screening | At screening
  Psychiatric screening will be assessed with the Mini-International Neuropsychiatric Interview
Beliefs about hypnosis | Before the procedure
  Beliefs about hypnosis will be assessed with an open-ended question "What are your beliefs about hypnosis?"
Expectancies about the study | Before the procedure
  Expectancies about the study will be assessed with an open-ended question "What are your expectancies about the study?"
Phenomenal control | During the procedure
  The phenomenal control will be assessed with the Phenomenological Control Scale.
Positive and negative affects | Beforethe procedure, During the procedure, direcly after the procedure, and after 3 months
  Positive and negative affects will be assessed with the Positive Affect and Negative Affect.
Absorption trait | Before the procedure
  The absorption trait will be assessed with the Tellegen Absorption Scale which consists of 34 true/false items, aiming to measure the absorption of a person, meaning the disposition for having episodes of a deep involvement that engage all the subject's resources (perceptual, imaginative, and cognitive). The total score range is from 0 to 34. The higher the score, the more one has a high propensity for absorption.
Dissociation trait | Before the procedure
  The dissociation trait will be assessed with the Dissociative Experience Scale. It is a self-reported questionnaire used to evaluate the presence, quantity, and type of dissociative experiences one might live in daily life. It consists of 28 items arranged on an analog scale (from 0 to 100% measuring the frequency of dissociative experiences), and the total score ranges from 0 to 100. There is a cutoff of 45 as a mean score to suggest a dissociative disorder. This questionnaire is not a diagnostic instrument; it is designed only for screening, but it can suggest that a specific clinical assessment is needed.
Anxiety state | Before the procedure and during the procedure
  Anxiety will be assessed with a numerical rating scale.
Absorption state | During the procedure
  Absorption will be assessed with a numerical rating scale.
Dissociation state | During the procedure
  Dissociation will be assessed with a numerical rating scale.
Alertness | During the procedure
  Alertness will be assessed with a numerical rating scale.
Time perception | During the procedure
  We will ask the participants how long they thought the intervention lasted.
Near Death Experience | During the procedure
  The near death experience will be assessed with the The Near-Death Experience Content (NDE-C) Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, Liège, Belgium